CLINICAL TRIAL: NCT06659731
Title: Pain Perception in Autism. Study Through Quantitative Sensory Testing and Psychophysiological Correlates
Brief Title: Quantitative Sensory Testing to Study Pain Perception in Autism
Acronym: PPiA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: id. 1043
Record Dates: First submitted 2024-10-14; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder (ASD); Pain Perception
Keywords: autism spectrum disorder (ASD); pain perception; somatosensory profile; children; QST
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD Group: Patients with ASD diagnosis according to DSM-V, between 5 and 17 years old
  Interventions: Other: Quantitative Sensory testing (QST); Other: EEG
- Control Group: Healthy participants, between 5 and 17 years old, without ASD diagnosis and withour neurological and psychiatric deseases
  Interventions: Other: Quantitative Sensory testing (QST); Other: EEG

INTERVENTIONS:
Other: Quantitative Sensory testing (QST) — The QST protocol (Rolke et al., 2006; Blankenburg et al., 2010), implies the administration of 7 short sensory test in order to measure up to 13 parameters, which can be grouped as follows: thermal detection thresholds for the perception of cold, warm and paradoxical heat sensations, thermal pain thresholds for cold and hot stimuli, mechanical detection thresholds for touch and vibration, mechanical pain thresholds and sensitivity for pinprick and blunt pressure, vibration detection threshold and pressure pain threshold.
Other: EEG — EEG recording at rest and while receiving heat stimuli to study cortical processing of salient thermal stimuli. Up to 30 painful thermal stimuli, will be delivered to the patients' hand dorsum in order to register contact heat evoked potentials (CHEPs).

SUMMARY:
This study aims at assess sensory perception, and pain perception, in neurodivergent children and adolescent in the autism spectrum. To achieve this goal, the quantitive sensory testing (QST), a controlled and replicable protocol, will be used, to assess perception in different sensory modalities: heat sensations, mechanical detection threshold and pain threshold. As secondary aim, the cortical processing of thermal painful stimuli will be collected through electroencephalography (EEG) in order to investigate if there are differences in the cortical processing of painful stimuli between clinical sample and control sample, and if it could be associated with differences in the subjective experience between the two groups. Finally, it will be explored the association between such differences, and indexes of psychopathology and dispositional measures.

DETAILED DESCRIPTION:
Study procedure imply the following steps: 1. Eligibility assessment according to inclusion and exclusion criteria. 2. Administration of questionnaires and scales for the characterization of clinical aspects of autism: Short sensory profile; The Autism Spectrum Quotient: Children's Version; Vineland Adaptive Behaviour Scales-Second Edition. The Vineland Adaptive Behaviour Scales-Second Edition; The Child Behavior Checklist (CBCL). 3. Administration of Quantitative Sensory Testing to study sensory thresholds and perception. 4. EEG recording at rest as well as while receiving heat stimuli to study cortical processing of salient thermal stimuli.

The QST protocol, implies the administration of 7 short sensory test in order to measure up to 13 parameters, which can be grouped as follows: thermal detection thresholds for the perception of cold, warm and paradoxical heat sensations, thermal pain thresholds for cold and hot stimuli, mechanical detection thresholds for touch and vibration, mechanical pain thresholds and sensitivity for pinprick and blunt pressure, vibration detection threshold and pressure pain threshold. Previous research with QST in neurodevelopmental disorders used modified version of the whole protocol, to make it suitable and tolerable for different clinical condition such as developmental delay including motor, communicative, and cognitive impairments. Thus, we will also administer the most suitable and tolerable version of the QST according to each patient condition and needs, for example we plan to reduce the number of stimuli for each stimulation side when needed, in order to reduce stimulus trial duration as well. The whole procedure will be implemented in a kids friendly environment, colourful and comfortable, and sensory stimuli will be adapted in order to avoid fearfulness of the stimuli, thus each stimulation will be presented as a game to be played with a specific animal, and each device and instrument will be covered with animals pictures according to the game it represents. Overall QST last about 1h 30 minutes, it will be divided in at least two sessions according to patients' needs.

The EEG recording consist in the cap montage at first, then a short accommodation with the sensory stimuli in order to find an intensity value for a moderate painful stimulus, to be used for the stimulation. After the preparation/accommodation, the eeg recording will start while a series, up to 30 thermal stimuli, will be delivered to the patients' hand dorsum. The whole eeg recording last about 30 minutes and it will be implemented in one session only.

ELIGIBILITY:
Inclusion Criteria for the clinical sample:

* Children and adolescent
* age between 5 and 17 years old
* Autism diagnosis according to DSM-V criteria

Inclusion Criteria for the control sample:

* healthy children and adolescent (without neurological, and psychiatric, diagnoses)
* age between 5 and 17 years old

Exclusion Criteria:

Comorbidities with (for the clinical sample) or diagnosis of (for the control sample):

* peripheral neuropaties;
* psychiatric diagnosis as psychosis,
* Tourette Syndrome,
* neurological diagnoses as epilepsy,
* sensory deficit or loss;
* genetic diseases

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescent between 5 and 17 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
EEG responses in the time domain | from the enrollment to the end of EEG recordin (approx. 3 days)
  ERPs amplitude (μV)
Cold detection threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (°C) at which a cold stimulus is perceived by each participant
Warm detection threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (°C) at which a warm stimulus is perceived by each participant
Cold pain threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (°C) at which a cold stimulus is perceived as painful by each participant
Warm pain threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (°C) at which a warm stimulus is perceived as painful by each participant
Mechanical detection threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (mN) at which a mechanical stimulus is perceived by each participant. It is a measure of touch perception
Mechanical pain threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (mN) at which a mechanical stimulus is perceived as painful by each participant.
Vibration detection threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (Hz) at which a vibratory stimulus is perceived by each participant.
Pressure pain threshold | from the enrollment to the end of QST administration (approx. 2 days)
  The minimum intensity value (N) at which a pressure stimulus is perceived as painful by each participant.
EEG responses in the time-frequency domain | from the enrollment to the end of QST administration (approx. 3 days)
  Power-spectrum of eeg responses

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS "E. Medea", Brindisi, BR, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoffman T, Bar-Shalita T, Granovsky Y, Gal E, Kalingel-Levi M, Dori Y, Buxbaum C, Yarovinsky N, Weissman-Fogel I. Indifference or hypersensitivity? Solving the riddle of the pain profile in individuals with autism. Pain. 2023 Apr 1;164(4):791-803. doi: 10.1097/j.pain.0000000000002767. Epub 2022 Aug 26. PMID 36730631
- [Background] Vaughan S, McGlone F, Poole H, Moore DJ. A Quantitative Sensory Testing Approach to Pain in Autism Spectrum Disorders. J Autism Dev Disord. 2020 May;50(5):1607-1620. doi: 10.1007/s10803-019-03918-0. PMID 30771132
- [Background] Chien YL, Chao CC, Wu SW, Hsueh HW, Chiu YN, Tsai WC, Gau SS, Hsieh ST. Small fiber pathology in autism and clinical implications. Neurology. 2020 Nov 10;95(19):e2697-e2706. doi: 10.1212/WNL.0000000000010932. Epub 2020 Oct 14. PMID 33055277
- [Background] Frundt O, Grashorn W, Schottle D, Peiker I, David N, Engel AK, Forkmann K, Wrobel N, Munchau A, Bingel U. Quantitative Sensory Testing in adults with Autism Spectrum Disorders. J Autism Dev Disord. 2017 Apr;47(4):1183-1192. doi: 10.1007/s10803-017-3041-4. PMID 28160223
- [Background] ZHANG Wenyun LX, YAO Junjie, YE Qian, PENG Weiwei. Abnormalities in pain sensitivity among individuals with autism spectrum disorder: Evidence from meta-analysis. Acta Psychologica Sinica 2021;53(6):613-628
- [Background] Proff I, Williams GL, Quadt L, Garfinkel SN. Sensory processing in autism across exteroceptive and interoceptive domains. Psychology & Neuroscience 2022;15(2):105
- [Background] Moore DJ. Acute pain experience in individuals with autism spectrum disorders: a review. Autism. 2015 May;19(4):387-99. doi: 10.1177/1362361314527839. Epub 2014 Mar 31. PMID 24687688
- [Derived] Nicolardi V, Fanizza I, Accogli G, Scoditti S, Trabacca A. Pain perception in autism. A study of sensory reactivity in children and adolescents with autism using quantitative sensory testing and psychophysiological correlates. Front Neurosci. 2025 May 1;19:1543538. doi: 10.3389/fnins.2025.1543538. eCollection 2025. PMID 40376609